CLINICAL TRIAL: NCT02885181
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Phase 2 Proof-of-Concept Study to Evaluate Safety, Tolerability, and Efficacy of GS-9876 in Subjects With Active Rheumatoid Arthritis on Background Therapy With Methotrexate
Brief Title: Safety, Tolerability, and Efficacy of GS-9876 in Participants With Active Rheumatoid Arthritis on Background Therapy With Methotrexate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-379-1582; 2016-001496-75 (EudraCT Number)
Record Dates: First submitted 2016-08-26; First posted 2016-08-31 (Estimated); Results first posted 2018-09-19 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — GLPG0634; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- GS-9876 - 30 mg (Experimental): GS-9876 30 mg + filgotinib placebo for 12 weeks
  Interventions: Drug: GS-9876; Drug: Filgotinib placebo; Drug: Methotrexate
- GS-9876 - 10 mg (Experimental): GS-9876 10 mg + filgotinib placebo for 12 weeks
  Interventions: Drug: GS-9876; Drug: Filgotinib placebo; Drug: Methotrexate
- Filgotinib (Experimental): Filgotinib + GS-9876 placebo for 12 weeks
  Interventions: Drug: Filgotinib; Drug: GS-9876 placebo; Drug: Methotrexate
- Placebo (Placebo Comparator): GS-9876 placebo + filgotinib placebo for 12 weeks
  Interventions: Drug: GS-9876 placebo; Drug: Filgotinib placebo; Drug: Methotrexate

INTERVENTIONS:
Drug: GS-9876 — One tablet administered orally once daily
  Arms: GS-9876 - 10 mg; GS-9876 - 30 mg
Drug: Filgotinib — Two tablets administered orally once daily
  Arms: Filgotinib
Drug: GS-9876 placebo — One tablet administered orally once daily
  Arms: Filgotinib; Placebo
Drug: Filgotinib placebo — Two tablets administered orally once daily
  Arms: GS-9876 - 10 mg; GS-9876 - 30 mg; Placebo
Drug: Methotrexate — Background therapy with methotrexate administered orally or parenterally once weekly

SUMMARY:
The primary objective of this study is to evaluate the effect of GS-9876 versus placebo for the treatment of signs and symptoms of rheumatoid arthritis (RA) in participants with active RA as measured by change from baseline in Disease Activity Score for 28 joint count using C-reactive protein (CRP) (DAS28 (CRP)) at Week 12.

ELIGIBILITY:
Key Inclusion Criteria:

* Active RA disease as defined by: a tender joint count (TJC) of ≥ 6 (out of 68), a swollen joint count (SJC) of ≥ 6 (out of 66) at screening and Day 1
* Inadequate response to treatment with oral or parenteral methotrexate (MTX) 7.5 to 25 mg/week continuously for at least 12 weeks
* No evidence of active or latent tuberculosis

Key Exclusion Criteria:

* Prior treatment with B-cell depleting agents (eg, rituximab), unless more than 6 months prior to the first dose of study drug and documented return of CD19+ cells at screening
* Prior treatment with any commercially available or investigational spleen tyrosine kinase (SYK) inhibitor
* Concurrent treatment with any other conventional synthetic DMARD (csDMARD) other than MTX and/or hydroxychloroquine (HCQ) (prior csDMARD treatment allowed if appropriate wash out as defined in the protocol)
* Concurrent treatment with any biological disease modifying anti-rheumatic drug (bDMARD)(prior bDMARD treatment allowed if appropriate wash out as defined in the protocol). Prior failure to treatment with bDMARDs is not an exclusion criterion.

Note: Other protocol defined Inclusion/ Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2016-09-21 (Actual); Primary Completion 2017-08-22 (Actual); Study Completion 2017-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (19):
- United States (9):
  - Omega Research Consultants, DeBary, Florida
  - Sarasota Arthritis Research Center, Sarasota, Florida
  - Medical Associates of North Georgia, Canton, Georgia
  - Center For Arthritis and Osteoporosis, Elizabethtown, Kentucky
  - Albuquerque Center For Rheumatology, Albuquerque, New Mexico
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Accurate Clinical Management - Najam, Houston, Texas
  - Accurate Clinical Research Inc., Stafford, Texas
  - Medical Center Research LLC, Webster, Texas
- Bulgaria (3):
  - MHAT-Plovdiv AD, Plovdiv
  - Umhat Kaspela, Plovdiv
  - NMTH Tsar Boris III, Sofia
- Czechia (2):
  - A-Shine s.r.o., Pilsen
  - Medical Plus, S.R.O., Uherské Hradiště
- LLC Arensia Exploratory Medicine, Tbilisi, Georgia
- ARENSIA Exploratory Medicine Phase I Unit, Republican Clinical Hospital, Chisinau, Moldova
- ClinicMed Badurski i wspolnicy Spolka Jawna, Bialystok, Poland
- Ukraine (2):
  - Kharkiv City Hospital 8, Kharkiv
  - Medical Center_Clinic of International Institute of clinical Studies, Kyiv

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States and Europe. The first participant was screened on 21 September 2016. The last study visit occurred on 20 September 2017.
Pre-assignment Details: 140 participants were screened.
Groups:
- GS-9876 30 mg: GS-9876 30 mg tablet orally once daily + filgotinib placebo 2 tablets orally once daily for 12 weeks and background therapy with methotrexate orally or parenterally once weekly
- GS-9876 10 mg: GS-9876 10 mg tablet orally once daily + filgotinib placebo 2 tablets orally once daily for 12 weeks and background therapy with methotrexate orally or parenterally once weekly
- Filgotinib: Filgotinib 2 x 100 mg tablets orally once daily + GS-9876 placebo tablet orally once daily for 12 weeks and background therapy with methotrexate orally or parenterally once weekly
- Placebo: GS-9876 placebo tablet orally once daily + filgotinib placebo 2 tablets orally once daily for 12 weeks and background therapy with methotrexate orally or parenterally once weekly
Period: Overall Study
Arm/Group | GS-9876 30 mg | GS-9876 10 mg | Filgotinib | Placebo
Started | 20 | 20 | 21 | 22
Completed | 20 | 19 | 21 | 19
Not Completed | 0 | 1 | 0 | 3
Not completed — Investigator's Discretion | 0 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who received at least 1 dose of study drug.
Groups:
- Filgotinib: Filgotinib 2 x 100 mg tablet orally once daily + GS-9876 placebo tablet orally once daily for 12 weeks and background therapy with methotrexate orally or parenterally once weekly
- Total: Total of all reporting groups
Arm/Group | GS-9876 30 mg | GS-9876 10 mg | Filgotinib | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 21 | 22 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (7.0) | 56 (11.4) | 53 (15.4) | 54 (10.9) | 55 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 17 | 21 | 69
  Male | 5 | 4 | 4 | 1 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2 | 0 | 4
  Not Hispanic or Latino | 19 | 19 | 19 | 22 | 79
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 2 | 4
  White | 20 | 17 | 21 | 19 | 77
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 00 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 8 | 8 | 9 | 33
  Czechia | 1 | 1 | 0 | 1 | 3
  Ukraine | 2 | 1 | 2 | 1 | 6
  Poland | 1 | 2 | 0 | 3 | 6
  Moldova | 3 | 5 | 6 | 4 | 18
  Georgia | 4 | 2 | 2 | 2 | 10
  Bulgaria | 1 | 1 | 3 | 2 | 7
Disease Activity Score 28 C-Reactive Protein (DAS28 CRP) [Mean (Standard Deviation); unit: units on a scale] — Disease Activity Score 28 C-Reactive Protein (DAS28 (CRP)) is a measure of the participant's disease activity calculated using the tender joint counts (28 joints), swollen joint counts (28 joints), participant's global assessment of disease activity (visual analog scale: 0 = no disease activity to 100 = maximum disease activity) and C-Reactive Protein (CRP) for a total possible score of 1 to 9.4.
  units on a scale | 5.78 (0.691) | 5.65 (0.941) | 6.09 (1.112) | 5.51 (1.003) | 5.75 (0.961)
Health Assessment Questionnaire Disease Index (HAQ-DI) [Mean (Standard Deviation); unit: units on a scale] — The Health Assessment Questionnaire - Disability Index (HAQ-DI) is a self-reported tool used to assess the ability to perform tasks in 8 functional categories: dressing and grooming, arising, eating, walking, hygiene, reach, grip, and common daily activities. Responses in each functional category were collected as 0 (without any difficulty) to 3 (unable to do a task in that area). The HAQ-DI score ranges from 0 (no disability) to 3 (completely disabled), when 6 or more categories are non-missing.
  units on a scale | 1.38 (0.650) | 1.47 (0.425) | 1.61 (0.591) | 1.51 (0.577) | 1.49 (0.563)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Disease Activity Score 28 C-Reactive Protein (DAS28 (CRP)) at Week 12
Description: Disease Activity Score 28 C-Reactive Protein (DAS28 (CRP)) is a measure of the participant's disease activity calculated using the tender joint counts (28 joints), swollen joint counts (28 joints), participant's global assessment of disease activity (visual analog scale: 0 = no disease activity to 100 = maximum disease activity) and C-Reactive Protein (CRP) for a total possible score of 1 to 9.4. Higher values indicate higher disease activity. A negative change from baseline indicates improvement.
Time Frame: Baseline; Week 12
Population: Participants in the Full Analysis Set (participants who received at least 1 dose of study drug) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GS-9876 30 mg | GS-9876 10 mg | Filgotinib | Placebo
Number analyzed (Participants) | 20 | 17 | 21 | 19
units on a scale | -1.26 (1.276) | -0.78 (1.119) | -2.46 (1.242) | -1.36 (1.044)
Statistical Analysis 1: Comparison: GS-9876 30 mg vs Placebo; Test type: Superiority; p = 0.978, Cochran-Mantel-Haenszel; Least Squares (LS) Means of Differences = 0.01, 95% CI 2-sided [- 0.74 to 0.76]
Statistical Analysis 2: Comparison: GS-9876 10 mg vs Placebo; Test type: Superiority; p = 0.300, Cochran-Mantel-Haenszel; LS Means of Differences = 0.40, 95% CI 2-sided [- 0.36 to 1.16]
Statistical Analysis 3: Comparison: Filgotinib vs Placebo; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel; LS Means of Differences = - 1.18, 95% CI 2-sided [- 1.92 to - 0.43]

2. Secondary Outcome: Percentage of Participants Who Achieved American College of Rheumatology (ACR)20 Improvement at Week 12
Description: American College of Rheumatology (ACR)20 response was defined as having ≥ 20% improvement from baseline in the number of tender and the number of swollen joints, and a 20% improvement in at least 3 of the following 5 criteria: Physician's Global Assessment of Disease Activity (PhGA), Participant's Global Assessment of Disease Activity (PtGA), Participant's pain assessment, Participant's assessment of physical function (HAQ-DI) score, and C-reactive protein (CRP).
Time Frame: Week 12
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Groups:
- GS-9876 - 10 mg: GS-9876 10 mg tablet orally once daily + Filgotinib placebo 2 tablets orally once daily for 12 weeks and background therapy with methotrexate orally or parenterally once weekly
Arm/Group | GS-9876 30 mg | GS-9876 - 10 mg | Filgotinib | Placebo
Number analyzed (Participants) | 20 | 20 | 21 | 22
percentage of participants | 35.0 | 25.0 | 81.0 | 40.9
Statistical Analysis 1: Comparison: GS-9876 30 mg vs Placebo; Test type: Superiority; p = 0.660, Cochran-Mantel-Haenszel; Difference in Response Rates = -5.9, 95% CI 2-sided [-36.0 to 24.0]
Statistical Analysis 2: Comparison: GS-9876 - 10 mg vs Placebo; Test type: Superiority; p = 0.277, Cochran-Mantel-Haenszel; Difference in Response Rates = -15.9, 95% CI 2-sided [-44.7 to 13.8]
Statistical Analysis 3: Comparison: Filgotinib vs Placebo; Test type: Superiority; p = 0.009, Cochran-Mantel-Haenszel; Difference in Response Rates = 40.0, 95% CI 2-sided [10.7 to 65.6]

3. Secondary Outcome: Percentage of Participants Who Achieved ACR50 Improvement at Week 12
Description: ACR50 response was defined as having ≥ 50% improvement from baseline in the number of tender and the number of swollen joints, and a 50% improvement in at least 3 of the following 5 criteria: PhGA, PtGA, Participant's pain assessment, HAQ-DI score, and CRP.
Time Frame: Week 12
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | GS-9876 30 mg | GS-9876 - 10 mg | Filgotinib | Placebo
Number analyzed (Participants) | 20 | 20 | 21 | 22
percentage of participants | 20.0 | 20.0 | 47.6 | 22.7
Statistical Analysis 1: Comparison: GS-9876 30 mg vs Placebo; Test type: Superiority; p = 0.853, Cochran-Mantel-Haenszel; Difference in Response Rates = -2.7, 95% CI 2-sided [-32.0 to 27.5]
Statistical Analysis 2: Comparison: GS-9876 - 10 mg vs Placebo; Test type: Superiority; p = 0.852, Cochran-Mantel-Haenszel; Difference in Response Rates = -2.7, 95% CI 2-sided [-32.0 to 27.5]
Statistical Analysis 3: Comparison: Filgotinib vs Placebo; Test type: Superiority; p = 0.092, Cochran-Mantel-Haenszel; Difference in Response Rates = 24.9, 95% CI 2-sided [-6.6 to 51.5]

4. Secondary Outcome: Percentage of Participants Who Achieved ACR70 Improvement at Week 12
Description: ACR70 response was defined as having ≥ 70% improvement from baseline in the number of tender and the number of swollen joints, and a 70% improvement in at least 3 of the following 5 criteria: PhGA, PtGA, Participant's pain assessment, HAQ-DI score, and CRP.
Time Frame: Week 12
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Groups:
- Filgotinib: Filgotinib 2 x 100 mg tablet orally once daily + GS-9876 placebo tablet orally once daily for 12 weeks Background therapy with methotrexate orally or parenterally once weekly
- Placebo: GS-9876 placebo tablet orally once daily + Filgotinib placebo 2 tablets orally once daily for 12 weeks Background therapy with methotrexate orally or parenterally once weekly
Arm/Group | GS-9876 30 mg | GS-9876 10 mg | Filgotinib | Placebo
Number analyzed (Participants) | 20 | 20 | 21 | 22
percentage of participants | 5.0 | 15.0 | 38.1 | 13.6
Statistical Analysis 1: Comparison: GS-9876 30 mg vs Placebo; Test type: Superiority; p = 0.360, Cochran-Mantel-Haenszel; Difference in Response Rates = -8.6, 95% CI 2-sided [-37.9 to 22.5]
Statistical Analysis 2: Comparison: GS-9876 10 mg vs Placebo; Test type: Superiority; p = 0.896, Cochran-Mantel-Haenszel; Difference in Response Rates = 1.4, 95% CI 2-sided [-28.0 to 31.7]
Statistical Analysis 3: Comparison: Filgotinib vs Placebo; Test type: Superiority; p = 0.072, Cochran-Mantel-Haenszel; Difference in Response Rates = 24.5, 95% CI 2-sided [-6.6 to 50.1]

5. Secondary Outcome: Change From Baseline in The Health Assessment Questionnaire - Disability Index (HAQ-DI) Score at Week 12
Description: The Health Assessment Questionnaire - Disability Index (HAQ-DI) is a self-reported tool used to assess the ability to perform tasks in 8 functional categories: dressing and grooming, arising, eating, walking, hygiene, reach, grip, and common daily activities. Responses in each functional category were collected as 0 (without any difficulty) to 3 (unable to do a task in that area). The HAQ-DI score ranges from 0 (no disability) to 3 (completely disabled), when 6 or more categories are non-missing.
Time Frame: Baseline; Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GS-9876 30 mg | GS-9876 10 mg | Filgotinib | Placebo
Number analyzed (Participants) | 20 | 19 | 21 | 19
units on a scale | -0.46 (0.480) | -0.18 (0.800) | -0.70 (0.649) | -0.39 (0.389)
Statistical Analysis 1: Comparison: GS-9876 30 mg vs Placebo; Test type: Superiority; p = 0.528, Cochran-Mantel-Haenszel; LS Means of Differences = -0.12, 95% CI 2-sided [-0.49 to 0.25]
Statistical Analysis 2: Comparison: GS-9876 10 mg vs Placebo; Test type: Superiority; p = 0.293, Cochran-Mantel-Haenszel; LS Means of Differences = 0.20, 95% CI 2-sided [-0.17 to 0.57]
Statistical Analysis 3: Comparison: Filgotinib vs Placebo; Test type: Superiority; p = 0.072, Cochran-Mantel-Haenszel; LS Means of Differences = -0.33, 95% CI 2-sided [-0.70 to 0.03]

ADVERSE EVENTS:
Time Frame: Up to 12 weeks + 30 days
Description: Safety Analysis Set
Arm/Group | GS-9876 30 mg | GS-9876 10 mg | Filgotinib | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/21 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/21 | 0/22
Other Adverse Events (participants affected / at risk) | 7/20 | 8/20 | 4/21 | 1/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GS-9876 30 mg (N=20) | GS-9876 10 mg (N=20) | Filgotinib (N=21) | Placebo (N=22)
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0
Meniere's disease (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 2 | 0 | 0 | 0
Hypermetropia (Eye disorders) | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 2 | 0
Condition aggravated (General disorders) | 0 | 2 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 1 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0
Liver function test increased (Investigations) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Amnesia (Nervous system disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (4):
  • Study Protocol: Original (2016-04-08): https://cdn.clinicaltrials.gov/large-docs/81/NCT02885181/Prot_000.pdf
  • Study Protocol: Amendment 1 (2016-06-27): https://cdn.clinicaltrials.gov/large-docs/81/NCT02885181/Prot_001.pdf
  • Study Protocol: Amendment 2 (2016-07-11): https://cdn.clinicaltrials.gov/large-docs/81/NCT02885181/Prot_002.pdf
  • Statistical Analysis Plan (2017-10-26): https://cdn.clinicaltrials.gov/large-docs/81/NCT02885181/SAP_003.pdf